CLINICAL TRIAL: NCT07378527
Title: A Phase II/III Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of ICP-332 in Moderate to Severe Chronic Spontaneous Urticaria Subjects Inadequately Controlled by Second Generation H1-antihistamines
Brief Title: Study of the Efficacy and Safety of ICP-332 in Participants With Chronic Spontaneous Urticaria
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00613
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Spontaneous Urticaria (CSU)
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ICP-332 dose A（Phase2） (Experimental): ICP-332 will be administered as tablet
  Interventions: Drug: ICP-332 Tablets
- ICP-332 dose B（Phase2） (Experimental): ICP-332 will be administered as tablet
  Interventions: Drug: ICP-332 Tablets
- ICP-332 dose C（Phase2） (Experimental): ICP-332 will be administered as tablet
  Interventions: Drug: ICP-332 Tablets
- Placebo（Phase2） (Placebo Comparator): ICP-332 Placebo will be administered as tablet
  Interventions: Drug: ICP-332 placebo Tablets
- ICP-332 dose A or dose B or dose C（Phase3） (Experimental): ICP-332 will be administered as tablet
  Interventions: Drug: ICP-332 Tablets
- Placebo（Phase3） (Placebo Comparator): ICP-332 Placebo will be administered as tablet
  Interventions: Drug: ICP-332 placebo Tablets

INTERVENTIONS:
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet for 12 weeks
  Arms: ICP-332 dose A（Phase2）; ICP-332 dose B（Phase2）; ICP-332 dose C（Phase2）
Drug: ICP-332 placebo Tablets — ICP-332 placebo will be administered as tablet for 12 weeks
  Arms: Placebo（Phase2）; Placebo（Phase3）
Drug: ICP-332 Tablets — ICP-332 will be administered as tablet for 24 weeks
  Arms: ICP-332 dose A or dose B or dose C（Phase3）

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ICP-332 in moderate to severe chronic spontaneous urticaria subjects inadequately controlled by second generation H1-antihistamines

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women aged 18 to 75 years.
* 2. Diagnosis of CSU inadequately controlled by second generation H1-antihistamines.
* 3. CSU duration for ≥ 6 months prior to randomization.
* 4. Before initiating any screening or study-specific procedures, the subject must voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. Having the other medical conditions related to CSU or other skin diseases/conditions.
* 2. Potential medical conditions or issues.
* 3. Pregnant female subjects or lactating female subjects.
* 4. The investigator determines that the subject is unsuitable for participating in this study for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Absolute change from baseline in UAS7 at Week 4. | 4 weeks
Phase 3: Absolute change from baseline in UAS7 at Week 12 | 12 weeks

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Bengbu Medical University First Affiliated Hospital, Bengbu, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - Xiangya hospital central south university, Changsha, Hunan
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Wuxi No. 2 People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shenyang Hospital of Integrated Traditional Chinese and Western Medicine （Shenyang Seventh People's Hospital）, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Provincial Hospital for Skin Disease, Shandong First Medical University, Jinan, Shandong
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Sichuan Academy of Medical Sciences&Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang